CLINICAL TRIAL: NCT05726890
Title: Early Childhood Insomnia: Underlying Mechanisms of Intervention Effects of the "Bedtime Checking" and the "Standard Checking" Methods
Brief Title: Examining the Effectiveness of Two Behavioral Interventions for Sleep Problems in Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Liat Tikotzky, Professor, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0276-22-SOR
Record Dates: First submitted 2023-01-23; First posted 2023-02-14 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Insomnia
Keywords: sleep; early childhood insomnia; infant; parent; behavioral sleep interventions
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bedtime checking (Experimental): The intervention is based on the principles of graduated extinction, defined as an "effective and recommended therapy in the treatment of bedtime problems and night-wakings" by the AASM. The basic guidelines for this intervention are: (1) When the infant shows tired signs, he/she should be put to bed awake; (2) parents should minimize their involvement after putting the infant to bed; (3) if the child protests/cries, the parent should check the infant's crib every few minutes (e.g., 5 minutes), briefly comfort the infant without taking him/her out of the crib, and help the infant resume a sleeping position/find sleep aids (e.g., pacifier); (4) disengage and leave the crib until the next visit, (5) In order to increase consistency, the same parent should implement the intervention.
  In the "bedtime checking" arm, parents will be instructed to implement the changes only at bedtime and will be asked to continue soothing their infant at night, as they normally do
  Interventions: Behavioral: bedtime intervention for early childhood insomnia
- standard checking (Active Comparator): Same as for "bedtime checking" at bedtime, but in the standard checking arm, parents apply the intervention guidelines also when the infant wakes up during the night.
  Interventions: Behavioral: bedtime and nighttime intervention for early childhood insomnia

INTERVENTIONS:
Behavioral: bedtime intervention for early childhood insomnia — The intervention focuses on providing parents with skills on how to modify and limit their sleep-related interactions with their infant at bedtime. These changes are expected to foster the infant's ability to fall asleep independently at bedtime. It is also expected that after 1-2 weeks, these changes would lead to self-soothing also during the night.
  Arms: bedtime checking
Behavioral: bedtime and nighttime intervention for early childhood insomnia — The intervention focuses on providing parents with skills on how to modify and limit their sleep-related interactions with their infant at bedtime and during the night. These changes are expected to foster the infant's ability to fall asleep independently at bedtime and to resume sleep independently during the night.
  Arms: standard checking

SUMMARY:
Behavioral insomnia of childhood affects 15-30% of infants. Behavioral interventions, based on limiting parent-child bedtime and nighttime interactions, are effective in significantly improving infant sleep problems. However, the implementation of these interventions frequently encompasses significant infant crying and parental distress that deter many parents. Research on gradual sleep interventions that involve a lower "dose" of parent-infant separation, and thus may be more acceptable by parents, has so far been sparse. The proposed study aims to advance research in this area through systematically studying the processes through which parent and infant factors impact treatment outcomes of a behavioral intervention method that involves parent-infant separation only at bedtime ("bedtime checking"), in comparison to an intervention that also directly targets night-wakings ("standard checking"/"graduated extinction").

DETAILED DESCRIPTION:
Early-childhood insomnia is very prevalent and is associated with negative child and family outcomes. Behavioral interventions, based on limiting parent-child nocturnal interactions, are effective in significantly improving infant sleep. However, these interventions frequently involve significant parent and infant distress that deter many parents. Research on gradual sleep interventions that involve a lower "dose" of parent-infant separation, and thus may be more accepted by many parents, has so far been sparse. Moreover, little scientific attention has been paid to factors that may underlie parental compliance with behavioral sleep interventions and treatment outcomes. Accordingly, the main aim of the proposed study is to study the processes through which parent and infant factors impact treatment adherence and outcomes of a behavioral intervention method that involves parent-infant separation only at bedtime ("bedtime checking"), compared to a method that also targets night-wakings ("standard checking").

The investigators will recruit 230 infants with early-childhood insomnia and their parents. Following a baseline assessment, infants will be randomly assigned to the "bedtime checking" intervention or to "standard checking". Sleep assessment will include actigraphy, videosomnography, and sleep logs. Parents will complete baseline procedures and questionnaires to assess intervention moderators (e.g., parental emotional distress, infant temperament). Daily diaries will be used to assess predictors/mediators of treatment adherence and outcomes (e.g., parental stress, couple support). Assessments will be conducted during the intervention, and at 4 weeks, 6-months and 12-months post-treatment.

The main hypotheses are: (1a) For parents who adhere to their intervention, the "standard checking" method will obtain sleep outcomes more quickly; (1b) The "bedtime checking" method will lead to higher parental adherence and lower attrition, compared to "standard checking"; (2) Significant interactions between baseline parent/infant risk characteristics and type of intervention would be found in the prediction of sleep outcomes; (3) In both groups, higher adherence to the intervention and better sleep outcomes will be predicted by: (i) lower parental stress, guilt, and distress attributions, and (ii) higher perceived couple support; By systematically studying, for the first time, the "bedtime checking" method (that probably will be more acceptable to many parents), compared to "standard checking", findings promise to shed light on theory-based mediators and moderators through which behavioral sleep interventions might exercise their benefits.

ELIGIBILITY:
Inclusion Criteria:

* Early-childhood insomnia according to DSM-5 criteria
* The parents wish to sleep independently from the child and would like the infant to need as little help as possible to fall asleep or stay asleep
* Two-parent, Hebrew-speaking families

Exclusion Criteria:

* Infants and parents with significant physiological sleep problems (e.g., sleep apnea)
* Infants and parents with any chronic health problems (based on self-report).

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in infant actigraphic number of night-wakings from baseline to 1-week and 2-week start of intervention | baseline and 1- and 2-week start of intervention
  Actigraphy, a wristwatch-like device, is a reliable method for measuring adults' and infants' sleep-wake patterns based on motility. The Sadeh validated scoring algorithms will be used to identify the number of night-wakings. Change will be examined from baseline to both 1-week and 2-week from start of intervention to examine the hypothesis that both interventions would lead to a reduction in the number of night-wakings but that standard checking would lead to a faster change than bedtime checking.
Change in parents' actigraphic number of night-wakings from baseline to 1-week and 2-week start of intervention | baseline and 1- and 2-week start of intervention
  Actigraphy, a wristwatch-like device, is a reliable method for measuring adults' and infants' sleep-wake patterns based on motility. The Sadeh validated scoring algorithms will be used to identify the number of night-wakings. Change will be examined from baseline to both 1-week and 2-week from start of intervention to examine the hypothesis that both interventions would lead to a reduction in the number of night-wakings but that standard checking would lead to a faster change than bedtime checking.
Change in infant actigraphic minutes awake during the night from baseline to 1-week and 2-week start of intervention | baseline and 1- and 2-week start of intervention
  Actigraphy, a wristwatch-like device, is a reliable method for measuring adults' and infants' sleep-wake patterns based on motility. The Sadeh validated scoring algorithms will be used to identify nocturnal wakefulness according to a 1-minute epoch interval. Change will be examined from baseline to both 1-week and 2-week from start of intervention to examine the hypothesis that both interventions would lead to a reduction in minutes awake, but that standard checking would lead to a faster change than bedtime checking.
Change in parents' actigraphic minutes awake during the night from baseline to 1-week and 2-week start of intervention | baseline and 1- and 2-week start of intervention
  Actigraphy, a wristwatch-like device, is a reliable method for measuring adults' and infants' sleep-wake patterns based on motility. The Sadeh validated scoring algorithms will be used to identify nocturnal wakefulness according to a 1-minute epoch interval. Change will be examined from baseline to both 1-week and 2-week from start of intervention to examine the hypothesis that both interventions would lead to a reduction in minutes awake, but that standard checking would lead to a faster change than bedtime checking.
Change in infant sleep logs' number of night-wakings from baseline to 1-week and 2-week start of intervention. | baseline and 1- and 2-week start of intervention
  Sleep logs have been validated relative to objective sleep measures, and they provide the parents' perspective on the infant and their own sleep. Parents will be asked to indicate each morning the number of times their infant woke up during the night. Change will be examined from baseline to both 1-week and 2-week from start of intervention to examine the hypothesis that both interventions would lead to a reduction in the number of night-wakings, but that standard checking would lead to a faster change than bedtime checking.
Change in parents' sleep logs' number of night-wakings from baseline to 1-week and 2-week start of intervention. | baseline and 1- and 2-week start of intervention
  Sleep logs have been validated relative to objective sleep measures, and they provide the parents' perspective on the infant and their own sleep. Parents will be asked to indicate each morning the number of times they woke up during the night. Change will be examined from baseline to both 1-week and 2-week from start of intervention to examine the hypothesis that both interventions would lead to a reduction in the number of night-wakings, but that standard checking would lead to a faster change than bedtime checking.
Change in infant sleep logs' minutes awake during the night from baseline to 1-week and 2-week start of intervention. | baseline and 1- and 2-week start of intervention
  Sleep logs have been validated relative to objective sleep measures, and they provide the parents' perspective on the infant and their own sleep. Parents will be asked to indicate each morning the length of time their infant was awake during the night. Change will be examined from baseline to both 1-week and 2-week from start of intervention to examine the hypothesis that both interventions would lead to a reduction in minutes awake, but that standard checking would lead to a faster change than bedtime checking.
Change in parents' sleep logs' minutes awake during the night from baseline to 1-week and 2-week start of intervention. | baseline and 1- and 2-week start of intervention
  Sleep logs have been validated relative to objective sleep measures, and they provide the parents' perspective on the infant and their own sleep. Parents will be asked to indicate each morning the length of time they were awake during the night. Change will be examined from baseline to both 1-week and 2-week from start of intervention to examine the hypothesis that both interventions would lead to a reduction in minutes awake, but that standard checking would lead to a faster change than bedtime checking.
Change in infant sleep logs' subjective sleep quality from baseline to 1-week and 2-week start of intervention. | baseline and 1- and 2-week start of intervention
  Parents will be asked to rate their infants' sleep quality on a scale ranging from 1 (bad) to 10 (excellent). Change will be examined from baseline to both 1-week and 2-week from start of intervention to examine the hypothesis that both interventions would lead to improved sleep quality, but that standard checking would lead to a faster change than bedtime checking.
Change in parents' sleep logs' subjective sleep quality from baseline to 1-week and 2-week start of intervention. | baseline and 1- and 2-week start of intervention
  Parents will be asked to rate their own sleep quality on a scale ranging from 1 (bad) to 10 (excellent). Change will be examined from baseline to both 1-week and 2-week from start of intervention to examine the hypothesis that both interventions would lead to improved sleep quality, but that standard checking would lead to a faster change than bedtime checking.
Attrition from intervention | baseline and 2-week start of intervention.
  The number of parents who drop out from the intervention. Change will be examined from baseline to end of the two-week intervention to examine the hypothesis that attrition from standard checking will be higher than from bedtime checking.

SECONDARY OUTCOMES:
Change in infant sleep logs' sleep latency from baseline to 2-week start of intervention | baseline and 2-week start of intervention.
  Parents will indicate how long it took their infant to fall asleep.
Change in infant actigraphic sleep duration from baseline to 2-week start of intervention | baseline and 2-week start of intervention.
  Actigraphy will be used to measure the number of true sleep minutes (excluding nighttime wakefulness) from sleep onset to morning awakenings.
Change in infant sleep-logs' sleep duration from baseline to 2-week start of intervention | baseline and 2-week start of intervention.
  Parents will indicate the number of hours their infant slept (excluding nighttime wakefulness).
Change in parents' actigraphic sleep duration from baseline to 2-week start of intervention | baseline and 2-week start of intervention.
  Actigraphy will be used to measure the number of true sleep minutes (excluding nighttime wakefulness) from sleep onset to morning awakenings.
Change in parents' sleep-logs' sleep duration from baseline to 2-week start of intervention | baseline and 2-week start of intervention.
  Parents will indicate the number of hours they slept (excluding nighttime wakefulness).
Change in infant actigraphic longest sleep period from baseline to 2-week start of intervention. | baseline and 2-week start of intervention.
  Actigraphy will be used to measure the longest sleep stretch during the night.
Change in parents' actigraphic longest sleep period from baseline to 2-week start of intervention. | baseline and 2-week start of intervention.
  Actigraphy will be used to measure the longest sleep stretch during the night.
Change in infant observed sleep latency from baseline to 2-week start of intervention. | baseline and 2-week start of intervention.
  Videosomnography will be used to assess the change in observed sleep latency. Scoring of sleep latency (a continuous variable) based on the video records will be based on established methods, developed by Thomas Anders. We consider these as secondary outcomes as we are not sure how many parents will be willing to use the cameras.
Change in infant observed number of night-wakings from baseline to 2-week start of intervention | baseline and 2-week start of intervention.
  Videosomnography will be used to assess the change in observed number of night-wakings. Scoring of the number of awakenings (a continuous variable) based on the videos, will be based on established methods, developed by Thomas Anders.
Change in infant observed minutes awake during the night from baseline to 2-week start of intervention | baseline and 2-week start of intervention.
  Videosomnography will be used to assess the change in observed minutes awake during the night. Scoring of minutes awake (a continuous variable) based on the video records will be based on established methods, developed by Thomas Anders.
Change in infant observed sleep duration from baseline to 2-week start of intervention. | baseline and 2-week start of intervention.
  Videosomnography will be used to assess the change in observed sleep duration. Scoring of sleep duration (a continuous variable) based on the video records will be based on established methods, developed by Thomas Anders.
Change in infant observed nocturnal self-soothing behavior (i.e., signaled night wakings out of total awakenings) from start of intervention to end of intervention. | First 3 days of intervention and last 3 days of intervention
  Videosomnography will be used to observe the change in the number of times the infant wakes up and signals out of total number of wakings.
Change in infant observed nocturnal self-soothing behavior from start of intervention to end of intervention. | First 3 days of intervention and last 3 days of intervention
  Videosomnography will be used to observe the change in the percent of infant self-soothing behaviors (e.g., looking for pacifier, use of comforting object) out of all soothing behaviors.
Adherence with intervention guidelines - interval from infant crying to parental approach | Measured daily during the two week intervention.
  Videosomnography will be used to observe the interval from the time of infant signaling to the time the parent approaches the crib.
Adherence with intervention guidelines - total time of parental presence in infant room | Measured daily during the two week intervention.
  Videosomnography will be used to observe the total time of parental presence in room as a response to infant cry.
Adherence with intervention guidelines - type of parental help. | Measured daily during the two week intervention.
  Videosomnography will be used to observe the type of parental response (e.g., short visit as guided, prolonged visit with active help).
Adherence with intervention guidelines based on daily logs. | Measured daily during the two week intervention.
  Parental daily logs will be employed to assess adherence using a scale from 1 (not at all) to 7 (very much). Parents in the bedtime checking group will report only in the evening. Parents in the standard checking group will report also in the morning regarding nighttime adherence.
Change in infant actigraphic number of night-wakings from baseline to 4 weeks post intervention and to 6 and 12 months post intervention. | baseline and 4 weeks, 6 months, 12 months post intervention.
  Actigraphy will be used to identify the number of night-wakings. Change will be examined from baseline to 4 weeks post intervention, and to 6 and 12 months post intervention.
Change in parent actigraphic number of night-wakings from baseline to 4 weeks post intervention and to 6 and 12 months post intervention. | baseline and 4 weeks, 6 months, 12 months post intervention.
  Actigraphy will be used to identify the number of night-wakings. Change will be examined from baseline to 4 weeks post intervention, and to 6 and 12 months post intervention.
Change in infant actigraphic minutes awake during the night from baseline to 4 weeks post intervention and to 6 and 12 months post intervention. | baseline and 4 weeks, 6 months, 12 months post intervention.
  Actigraphy will be used to identify minutes awake during the night. Change will be examined from baseline to 4 weeks post intervention, and to 6 and 12 months post intervention.
Change in parent actigraphic minutes awake during the night from baseline to 4 weeks post intervention and to 6 and 12 months post intervention. | baseline and 4 weeks, 6 months, 12 months post intervention.
  Actigraphy will be used to identify minutes awake during the night. Change will be examined from baseline to 4 weeks post intervention, and to 6 and 12 months post intervention.
Change in infant daily logs' number of night-wakings from baseline to 4 weeks post intervention and to 6 and 12 months post intervention. | baseline and 4 weeks, 6 months, 12 months post intervention.
  Parents will use sleep logs to indicate each morning the number of times their infant woke up during the night. Change will be examined from baseline to 4 weeks post intervention, and to 6 and 12 months post intervention.
Change in parent daily logs' number of night-wakings from baseline to 4 weeks post intervention and to 6 and 12 months post intervention. | baseline and 4 weeks, 6 months, 12 months post intervention.
  Parents will use sleep logs to indicate each morning the number of times they woke up during the night. Change will be examined from baseline to 4 weeks post intervention, and to 6 and 12 months post intervention.
Change in infant daily logs' minutes awake during the night from baseline to 4 weeks post intervention and to 6 and 12 months post intervention. | baseline and 4 weeks, 6 months, 12 months post intervention.
  Parents will use sleep logs to indicate each morning how many minutes their infant was awake during the night. Change will be examined from baseline to 4 weeks post intervention, and to 6 and 12 months post intervention.
Change in parent daily logs' minutes awake during the night from baseline to 4 weeks post intervention and to 6 and 12 months post intervention. | baseline and 4 weeks, 6 months, 12 months post intervention.
  Parents will use sleep logs to indicate each morning how many minutes they were awake during the night. Change will be examined from baseline to 4 weeks post intervention, and to 6 and 12 months post intervention.
Change in parents' subjective rating of the infant's sleep problem from baseline to 4 weeks post intervention and to 6 and 12 months post intervention. | baseline and 4 weeks, 6 months, 12 months post intervention.
  One item from the Brief Infant Sleep Questionnaire will be used to examine change in parental perception of their infant's sleep problems: "Do you consider your child's sleep as a problem?":1= not at all to 5 = very much

CONTACTS AND LOCATIONS:
Overall Officials: Liat Tikotzky, PhD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Ben-Gurion University of the Negev, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No
Individual data will be kept confidential.

REFERENCES:
- [Background] Mindell JA, Kuhn B, Lewin DS, Meltzer LJ, Sadeh A; American Academy of Sleep Medicine. Behavioral treatment of bedtime problems and night wakings in infants and young children. Sleep. 2006 Oct;29(10):1263-76. PMID 17068979
- [Background] Tikotzky L, Sadeh A. The role of cognitive-behavioral therapy in behavioral childhood insomnia. Sleep Med. 2010 Aug;11(7):686-91. doi: 10.1016/j.sleep.2009.11.017. PMID 20620108
- [Background] Meltzer LJ, Mindell JA. Systematic review and meta-analysis of behavioral interventions for pediatric insomnia. J Pediatr Psychol. 2014 Sep;39(8):932-48. doi: 10.1093/jpepsy/jsu041. Epub 2014 Jun 19. PMID 24947271
- [Background] Sadeh A. Assessment of intervention for infant night waking: parental reports and activity-based home monitoring. J Consult Clin Psychol. 1994 Feb;62(1):63-8. doi: 10.1037//0022-006x.62.1.63. PMID 8034831
- [Background] Eckerberg B. Treatment of sleep problems in families with young children: effects of treatment on family well-being. Acta Paediatr. 2004 Jan;93(1):126-34. doi: 10.1080/08035250310007754. PMID 14989452
- [Background] Kahn M, Juda-Hanael M, Livne-Karp E, Tikotzky L, Anders TF, Sadeh A. Behavioral interventions for pediatric insomnia: one treatment may not fit all. Sleep. 2020 Apr 15;43(4):zsz268. doi: 10.1093/sleep/zsz268. PMID 31676910
- [Background] Gradisar M, Jackson K, Spurrier NJ, Gibson J, Whitham J, Williams AS, Dolby R, Kennaway DJ. Behavioral Interventions for Infant Sleep Problems: A Randomized Controlled Trial. Pediatrics. 2016 Jun;137(6):e20151486. doi: 10.1542/peds.2015-1486. PMID 27221288